CLINICAL TRIAL: NCT04475328
Title: Efficacy and Safety of AngongNiuhuang Pill in Patients With Acute Ischemic Stroke
Brief Title: Efficacy and Safety of AngongNiuhuang Pill in Patients With Acute Ischemic Stroke (ANGONG TRIAL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bin Peng, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUMCH-AGNH2020
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; AngongNiuhuang Pill
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AngongNiuhuang (Experimental): Drugs : AngongNiuhuang pill. The other treatments will provided according to guidelines for standard treatment of acute ischemic stroke.
  Interventions: Drug: AngongNiuhuang pill; Other: Standard treatment
- Placebo of AngongNiuhuang (Placebo Comparator): Drugs : Placebo of AngongNiuhuang pill. The other treatments will provided according to guidelines for standard treatment of acute ischemic stroke.
  Interventions: Drug: Placebo of AngongNiuhuang pill; Other: Standard treatment

INTERVENTIONS:
Drug: AngongNiuhuang pill — This group will receive AngongNiuhuang pill 1pill qd/day for 5-day.
  Other Names: Angong Niuhuang Wan
  Arms: AngongNiuhuang
Drug: Placebo of AngongNiuhuang pill — This group will receive placebo of AngongNiuhuang pill 1pill qd/day for 5-day.
  Other Names: Placebo of Angong Niuhuang Wan
  Arms: Placebo of AngongNiuhuang
Other: Standard treatment — The other treatments according to guidelines for standard treatment of acute ischemic stroke

SUMMARY:
AngongNiuhuang pill has obvious effects on the cardiovascular and cerebrovascular diseases. Pharmacological experiments confirmed that AngongNiuhuang pill can protect blood-brain barrier, inhibit capillary permeability, improve the tolerance of cerebral ischemia and hypoxia, reduce oxidative stress injury, thus protecting brain tissue. Clinical studies have also confirmed that AngongNiuhuang pill can increase the GCS score, reduce coma, improve nerve function defect and promote nerve function recovery. The primary purpose of this trial was to evaluate the difference in the volume of cerebral infarction and cerebral edema between Angong Niuhuang pill and placebo in patients with ischemic stroke at 14 days compared with the baseline.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, double-blinded, placebo parallel controlled, multicenter trial. Patients who met the inclusion and exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive AngongNiuhuang pill 1pill qd/day for 5-day; 2) the other group will receive Placebo of AngongNiuhuang pill 1pill qd/day for 5-day. The primary purpose of this trial was to evaluate the difference in the volume of cerebral infarction and cerebral edema between Angong Niuhuang pill and placebo in patients with ischemic stroke at 14 days compared with the baseline. The study was consisted of six visits, including the day of randomization, 2 days, 3-6 days, 7 days (the endap time of the therapy), 14 days, and 90 days (the endap time of the follow-up). Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment neurological function rating scale will be recorded during the program. The period of the trial is from August 2020 to October 2021, and 120 subjects are planned to be recruited from 10 centers in China. All the related investigative organizations and individuals will obey the Declaration of Helsinki and Chinese Guard-cell protoplast (GCP) standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participates aged 40-80 years.
2. Diagnosis with acute ischemic stroke.
3. Diagnosis with acute cerebral infarctions of internal carotid artery system.
4. 10≤ Baseline NIHSS <20.
5. Time of onset ≤36h.
6. Provision of informed consent.

Exclusion Criteria:

1. Not suitable for taking this medicine according to the judgement of consulting traditional Chinese medical doctor.
2. Suffering from intracranial tumors, encephalitis, subarachnoid hemorrhage and other brain organic diseases.
3. Patients with hemorrhagic transformation after cerebral infarction.
4. Received or planned to receive endovascular treatment, including thrombectomy, ultra early thrombectomy and stenting.
5. Received or planned to receive decompression craniectomy.
6. With mRS score >1 before onset of this episode.
7. Participates who cannot tolerate the MRI scans, such as Using a pacemaker or automatic defibrillator or having claustrophobia.
8. With thrombocytopenia (<100 x10^9/L), hematologic diseases or other systemic bleeding tendency.
9. With Alanine transaminase or Aspartate aminotransferase >1.5 times than normal upper limit or Creatinine >1.5 times than normal upper limit.
10. Allergic to ingredients of AngongNiuhuang pill.
11. Received AngongNiuhuang pill within 1 month.
12. Participates who plan to become pregnant within 3 months, or women of childbearing age with negative pregnancy test but refuse to accept contraception; during pregnancy or lactation.
13. Participates in other clinical trials within 30 days before randomization or currently involved in other clinical trails.
14. Participates with a life expectancy less than 3 months.
15. Incapable to follow this study due to mental illness, cognitive or emotional disorders.
16. Participates are not eligible for this clinical trial as evaluated by the investigators.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Cerebral infarction volume | 14 days
  Changes in cerebral infarction volume on Day 14 of the treatment from baseline.
Cerebral edema volume | 14 days
  Changes in cerebral edema volume on Day 14 of the treatment from baseline.
The proportion of the patients with Severity Adverse Events within 90 days of the treatment. | 90 days
  Severity Adverse Events

SECONDARY OUTCOMES:
Cerebral infarction volume | 90 days
  Changes in cerebral infarction volume on Day 90 of the treatment from baseline.
Cerebral edema volume | 90 days
  Changes in cerebral edema volume on Day 90 of the treatment from baseline.
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 2 point on the Day 14 and 90 of treatment. | 14 days, 90 days
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome.
Changes in NIHSS score on Day 14 and 90 of the treatment from baseline. | 14 days, 90 days
  The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Changes in Glasgow Coma Score (GCS) on the Day 7 and 14 of the treatment from baseline. | 7 days, 14 days
  We will use the GCS score to evaluate the degree of coma. The GCS have three domain items (open-eye response, speech response, and movement). The maximum possible score is 15, with the minimum score being a 3.
Changes of biomarker (hs-CRP) | 7 days
  Evaluation of the change in hs-CRP on Day 7 of the treatment.
Changes of biomarker (MMP-9) | 7 days
  Evaluation of the change in MMP-9 on Day 7 of the treatment.
Changes of biomarker (S-100B) | 7 days
  Evaluation of the change in S-100B on Day 7 of the treatment.
Changes of biomarker (NSE) | 7 days
  Evaluation of the change in NSE on Day 7 of the treatment.
The proportion of the patients with Severity Adverse Events within 7 days of the treatment. | 7 days
  Severity Adverse Events
Changes in toxicology index including mercury and arsenic on Day 7 of the treatment. | 7 days
  toxicology index
The proportion of the patients with Adverse Events within 7 and 90 days of the treatment. | 7 days, 90 days
  Adverse Events
The proportion of the patients with All-cause mortality within 7 and 90 days of the treatment. | 7 days, 90 days
  All-cause mortality
The proportion of the patients with Combined vascular events within 7 and 90 days of the treatment. | 7 days, 90 days
  Combined vascular events

CONTACTS AND LOCATIONS:
Overall Officials: Bin Peng, MD, Principal Investigator — Peking Union Medical College Hosptial, Chinese Academy of Medical Sciences
Locations (1):
- Department of Neurology,Peking Union Medical College Hospital,Shuaifuyuan 1,Dong Cheng District. Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Wang A, Shi L, Liu Q, Guo X, Liu K, Wang X, Li J, Zhu J, Wu Q, Yang Q, Zhuang X, You H, Feng F, Luo Y, Li H, Ni J, Peng B. Safety and efficacy of Angong Niuhuang Pills in patients with moderate-to-severe acute ischemic stroke (ANGONG TRIAL): A randomized double-blind placebo-controlled pilot clinical trial. Chin Med J (Engl). 2025 Mar 5;138(5):579-588. doi: 10.1097/CM9.0000000000003133. Epub 2024 Nov 6. PMID 39501831